CLINICAL TRIAL: NCT01295281
Title: A Prospective, Randomized, Cross-over Study - Evaluation of a New Catheter Material for Intermittent Catheterization
Brief Title: Evaluation of a New Catheter Material for Intermittent Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LOF-0018
Record Dates: First submitted 2011-01-21; First posted 2011-02-14 (Estimated); Results first posted 2014-03-03 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Catheterization (Clean, Intermittent Urinary Catheterization)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LoFric POBE 2.0 - PVC (Experimental): First period (7 days) use of LoFric POBE 2.0 followed by second period (7 days) use of LoFric PVC
  Interventions: Device: LoFric POBE 2.0; Device: LoFric PVC
- LoFric PVC - POBE 2.0 (Experimental): First period (7 days) use of LoFric PVC followed by second period (7 days) use of LoFric POBE 2.0.
  Interventions: Device: LoFric POBE 2.0; Device: LoFric PVC

INTERVENTIONS:
Device: LoFric POBE 2.0 — To be used at least twice daily, during 7 days. Treatment period 1 and 2 last 7 days, respectively.
Device: LoFric PVC — To be used at least twice daily, during 7 days. Treatment period 1 and 2 last 7 days, respectively.

SUMMARY:
The hypothesis to be investigated is if the tolerability of intermittent catheterization with Polyolefin Based Elastomer (POBE) 2.0 and Polyvinyl Chloride (PVC) is clinically equal - i.e. clinically non-inferior when using POBE 2.0 compared to PVC.

Secondary objectives are to evaluate the safety and the subject's perception associated with the use of the catheters, assessed by the recording of adverse events and the ease of handling by means of a subjective assessment scale.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Males, aged 18 years and over
* Maintained urethra sensibility
* Practice intermittent self-catheterization at least 2 times daily
* Using catheters in the length of 40 cm and size charrière (Ch) 12 or Ch 14
* Experienced practitioners of intermittent self-catheterization defined as a minimum of three months on therapy
* Experience of using LoFric catheter within the last 12 months prior to study entry
* Adults able to read, write and understand information given to them regarding the study

Exclusion Criteria:

* Ongoing, symptomatic urinary tract infection (UTI) at enrolment as judged by investigator
* Known urethral stricture at enrolment as judged by investigator
* Involvement in the planning and/or conduct of the study (applies to both Astra Tech staff or staff at the study site)
* Previous enrolment or randomisation of treatment in the present study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Johansson, Urotherapist, Principal Investigator — Kärnsjukhuset Skövde
Locations (6):
- Sweden (6):
  - Kirurg och Urologmottagningen, Alingsås lasarett, Alingsås
  - Urologcentrum, Borås
  - Kirurg- och urologmottagningen, Gävle Sjukhus, Gävle
  - Urologmottagningen, Lundby Sjukhus, Gothenburg
  - Uroterapimottagningen Kärnsjukhuset Skövde, Skövde
  - Urologmottagningen Uddevalla sjukhus, Uddevalla

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 107 subjects were enrolled in the study but 105 started treatment, i.e. two subjects dropped out before start of treatment. Both these subjects missed to fulfil all inclusion criteria.
  53 subjects started using LoFric Polyolefin Based Elastomer (POBE) 2.0 and 52 subjects started using LoFric Polyvinyl Chloride (PVC).
Period: First Intervention (7 Days)
Arm/Group | LoFric POBE 2.0 - PVC | LoFric PVC - POBE 2.0
Started | 53 | 52
Completed | 53 | 51
Not Completed | 0 | 1
Not completed — Death | 0 | 1
Period: Second Intervention (7days)
Arm/Group | LoFric POBE 2.0 - PVC | LoFric PVC - POBE 2.0
Started | 53 | 51
Completed | 53 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LoFric POBE 2.0 - PVC | LoFric PVC - POBE 2.0 | Total
Number analyzed (Participants) | 53 | 52 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (10) | 72 (10) | 72 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 53 | 52 | 105
Region of Enrollment [Number; unit: participants]
  Sweden | 53 | 52 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Discomfort
Description: The primary objective of this study is to compare the subject's tolerability, with regards to perceived discomfort, when using two different urinary catheters. Perception of discomfort (yes/ no) will be assessed in patient questionnaire for each subject. The frequency of discomfort will be compared between the treatments.
Time Frame: At 7 and 14 days after randomization, respectively
Population: Since the study is cross-over, all (104) subjects evaluated both LoFric POBE 2.0 and LoFric PVC. To be able to group and describe the results the "Arm/Group Titles" are renamed in this section to "LoFric POBE 2.0" and "LoFric PVC" respectively. Each Arm/Group describing the outcome for all 104 subjects (ITT analysis set).
Measure: Number; unit: participants
Groups:
- LoFric POBE 2.0: Single use LoFric POBE 2.0 catheters were used for intermittent catheterization at least twice daily for seven days. Catheterization was performed by the subjects themselves in a home setting.
- LoFric PVC: Single use LoFric PVC catheters were used for intermittent catheterization at least twice daily for seven days. Catheterization was performed by the subjects themselves in a home setting.
Arm/Group | LoFric POBE 2.0 | LoFric PVC
Number analyzed (Participants) | 104 | 104
participants | 15 | 29
Statistical Analysis 1: Comparison: LoFric POBE 2.0 vs LoFric PVC; The size of the target population was estimated by calculating 95% Confidence Interval (CI) of a possible difference between the two catheter types. The width of the interval was decided on the proportion of patients who would prefer one or the other catheter. Max width was seen when both proportions were 0.5. A total of 90 evaluable subjects limited the maximum width to 0.41, which was considered narrow enough from a scientific point of view, why this sample size was used in the study; Test type: Non-Inferiority or Equivalence — Two catheters were tested regarding subjects' perception when using them, in a cross over design. After using each catheter for 1 week the subjects were asked: "Do you experience discomfort when using your catheter"?, and the subjects were supposed to answer "Yes" or "No". The hypothesis to be investigated was that the tolerability/perception was about the same for each type of catheter, i.e. the POBE 2.0 should be non-inferior compared to PVC. H0: p(disc. POBE - Yes) = p(disc. PVC - Yes); p = 0.0066, McNemar

2. Secondary Outcome: Perception of Pain
Description: To compare subject's tolerability with regards to perceived pain, when using two different urinary catheters; PVC vs. POBE 2.0. Assessed in patient questionnaire for each subject. A 5-graded scale will be used to determine the perception and the severity of each variable. The difference between the treatments will be calculated for each subject.
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

3. Secondary Outcome: Perception of Burning Sensation
Description: To compare subject's tolerability with regards to perceived burning sensation, when using two different urinary catheters; PVC vs. POBE 2.0. Assessed in patient questionnaire for each subject. A 5-graded scale will be used to determine the perception and the severity of each variable. The difference between the treatments will be calculated for each subject.
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

4. Secondary Outcome: Presence of Bleeding
Description: To compare subject's tolerability with regards to presence of bleeding, when using two different urinary catheters; PVC vs. POBE 2.0. Assessed in patient questionnaire for each subject. A 5-graded scale will be used to determine the perception and the severity of each variable. The difference between the treatments will be calculated for each subject.
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

5. Secondary Outcome: Perception of "Other Discomfort"
Description: To compare subject's tolerability with regards to perceived "other discomfort", when using two different urinary catheters; PVC vs. POBE 2.0. Frequency of "other discomfort" (yes/ no) will be assessed in patient questionnaire. The frequency of "other discomfort" will be compared between the treatments. "Other discomfort" will be further specified using 5-graded scale (as for the other variables on the 5-graded scale the difference between the treatments will be calculated for each subject).
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

6. Secondary Outcome: Perception of Stiffness/ Rigidity
Description: To evaluate subject perception related to the physical properties of the catheter, when practising intermittent self catheterization with urinary catheters; PVC vs. POBE 2.0. Assessed in patient questionnaire for each subject. A 5-graded scale will be used to determine the perception and the severity of each variable. The difference between the treatments will be calculated for each subject.
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

7. Secondary Outcome: Perception of Catheter Eyes
Description: as for outcome 6
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

8. Secondary Outcome: Perception of Catheter Adherence
Description: as for outcome 6
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

9. Secondary Outcome: Perception of Catheter Tip
Description: as for outcome 6
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

10. Secondary Outcome: Perception of Slipperiness
Description: To evaluate subject perception related to the properties of the catheter's coating/surface, when practising intermittent self catheterization with urinary catheters; PVC vs. POBE 2.0. Assessed in patient questionnaire for each subject. A 5-graded scale will be used to determine the perception and the severity of each variable. The difference between the treatments will be calculated for each subject.
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

11. Secondary Outcome: Perception of Smoothness
Description: as for outcome 10
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

12. Secondary Outcome: Perception of Resistance
Description: as for outcome 10
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

13. Secondary Outcome: Perception of Discomfort Due to Other Causes
Description: To compare subject's tolerability with regards to perceived discomfort due to other causes, when using two different urinary catheters 2.0. Frequency of discomfort due to other causes (yes/ no) will be assessed in patient questionnaire. The frequency of discomfort due to other causes will be compared between the treatments. Discomfort due to other causes will be further specified using 5-graded scale (as for the other variables on the 5-graded scale the difference between the treatments will be calculated for each subject).
Time Frame: At 7 and 14 days after randomization, respectively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent until End of Study, up to 14 days.
Arm/Group | LoFric POBE 2.0 | LoFric PVC
Serious Adverse Events (participants affected / at risk) | 1/104 | 2/105
Other Adverse Events (participants affected / at risk) | 14/104 | 26/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LoFric POBE 2.0 (N=104) | LoFric PVC (N=105)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Abnormal potassium level during planned cytostatic treatment (Surgical and medical procedures) | 1 (1) | 0 (0)
Snakebite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LoFric POBE 2.0 (N=104) | LoFric PVC (N=105)
Bleeding in connection to catheterization (Renal and urinary disorders) | 3 | 7
Burning sensation in connection to catheterization (Renal and urinary disorders) | 11 | 21
Pain in connection to catheterization (Renal and urinary disorders) | 14 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days